CLINICAL TRIAL: NCT01655771
Title: A Phase 1, Open-Label, Single-Dose, Parallel-Group Study to Assess the Safety, Tolerability, and Pharmacokinetics of TD-1211 Administered Orally to Elderly and Young Healthy Subjects
Brief Title: TD-1211 Single-Dose Study in Elderly and Young Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0083
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Constipation
Keywords: Opioid induced constipation; Constipation
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly (Experimental): TD-1211 Dose 1
  Interventions: Drug: TD-1211 Dose 1
- Younger (Experimental): TD-1211 Dose 2
  Interventions: Drug: TD-1211 Dose 2

INTERVENTIONS:
Drug: TD-1211 Dose 1
  Arms: Elderly
Drug: TD-1211 Dose 2
  Arms: Younger

SUMMARY:
The purpose of this study is to measure the way in which TD-1211 is absorbed and eliminated by the body and to evaluate whether it is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* For the elderly cohort, nonsmoking 65 to 85 years, inclusive. For the young cohort, nonsmoking 18 to 45 years, inclusive.
* Body mass index (BMI) should be 18 to 36 kg/m2, inclusive.
* At screening, sitting or supine heart rate of 50 to 100 beats per minute and sitting or supine systolic and diastolic blood pressure of 90 to 150 mm Hg and 50 to 90 mm Hg, respectively (2 of 3 measurements)
* Subjects with mild, chronic, stable disease (e.g., controlled hypertension, non-insulin-dependent diabetes, arthritis) may be enrolled if deemed medically acceptable by the investigator
* Negative for hepatitis B virus, hepatitis C virus, and human immunodeficiency virus antibody within the last 3 months
* No clinically relevant abnormalities in laboratory evaluations

Exclusion Criteria:

* History or presence of clinically significant respiratory, gastrointestinal, renal, hepatic, endocrine, hematological, neurological (including chronic headache, current or prior psychiatric disease/condition, stroke), cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, or dermatological disorders. Subjects with mild, chronic, stable disease (e.g., controlled hypertension, controlled hypercholesterolemia, non insulin-dependent diabetes, osteoarthritis) may be enrolled if condition is well controlled and not anticipated to interfere with the objectives of the study.
* Any clinically significant abnormal ECG (electrocardiogram).
* Participation in another clinical trial of an investigational drug or medical device within 60 days.
* Donation of ≥500 mL blood, or equivalent, within 8 weeks prior to admission day.
* Any other condition that, in the opinion of the investigator, would confound or interfere with evaluation of safety, tolerability, or PK of the investigational drug or prevent compliance with the study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-96 hours
AUCt | Based on samples collected 0-96 hours
AUCinf | Based on samples collected 0-96 hours

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events | Days 1-14
Number patients with abnormal vital sign measurements | Days 1-5
Number of patients with abnormal clinical laboratory results | Days 1-5
Number of patients with abnormal corrected QTc interval | Days 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- ICON Development Solutions, San Antonio, Texas, United States